CLINICAL TRIAL: NCT04296461
Title: Phase 1 Open-Label, Dose-Escalation Study to Evaluate the Safety and Tolerability of Welgenaleucel (UWC19) in Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: Study of Welgenaleucel (UWC19) in Patients With Relapsed or Refractory B-cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UWELL Biopharma (Industry)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UBP-PCL-P01-3002-01
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-03

CONDITIONS: B-cell Non-Hodgkin Lymphoma
Keywords: CD19; non-Hodgkin lymphoma; CAR-T cells
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: A standard 3+3 trial design will be used Welgenaleucel(UWC19) dose escalation cohorts. The planned dose escalation cohort levels for Welgenaleucel (UWC19) are 4, 8, 12, 16 and 20 x10^6 CAR-T cells/kg.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Welgenaleucel (UWC19) (Experimental): Part I The safety and efficacy of Welgenaleucel (UWC19) will be evaluated in a standard 3+3 dose escalation approach.The planned dose escalation cohort levels for Welgenaleucel (UWC19) are 4, 8, 12, 16 and 20 x10^6 CAR-T cells/kg administered intravenously once.
  Interventions: Genetic: Welgenaleucel

INTERVENTIONS:
Genetic: Welgenaleucel — Welgenaleucel (UWC19) is a CD19-directed immunotherapy consisting of autologous T cells, which is reprogrammed to target cells that express CD19.
  Other Names: UWC19

SUMMARY:
This is an open-label, single-center Phase 1/2 study with a dose-escalation phase (Part 1) and a cohort expansion phase (Part 2) in patients with relapsed or refractory (R/R) B-cell non-Hodgkin lymphoma (B-NHL).

ELIGIBILITY:
Inclusion Criteria:

Have a primary diagnosis of B cell non-Hodgkin lymphoma

- Histologically confirmed: Diffuse Large B Cell Lymphoma (DLBCL), Primary Mediastinal Large B Cell Lymphoma (PMBCL), Transformation Follicular Lymphoma (TFL), High grade B-cell Lymphoma (HGBCL), Mantle cell Lymphoma (MANT), Burkitt Lymphoma (BURK), Lymphoblastic Lymphoma

* Chemotherapy-refractory disease, defined as one of more of the following No response to last line of therapy OR Refractory post-autologous stem cell transplant (ASCT)
* Individuals must have received adequate prior therapy including at a minimum:

anti-CD20 monoclonal antibody unless investigator determines that tumor is CD20-negative and an anthracycline containing chemotherapy regimen for individual with transformed FL must have chemorefractory disease after transformation to DLBCL.

* No active infection of HIV, HTLV and Syphilis
* Adequate renal function
* Adequate hepatic function
* Adequate cardiac function
* Adequate venous access for apheresis, and no other contraindications for leukapheresis
* Voluntary informed consent is given.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Received allogeneic Hematopoietic Stem Cell Transplantation (alloHSCT)
* Body weight less than 30 kg
* Pregnant or lactating women.
* Uncontrolled active infection.
* History of hepatitis B or hepatitis C infection.
* Previously treatment with any gene therapy products or cell therapy product in past 28 days.
* HIV infection.
* Lymphoma with central nervous system (CNS) involvement
* Have autoimmune disorders
* Have active infection or inflammatory disorders
* Prescreening test results in expansion rate less than 5 folds
* An allergy to gentamycin and/or streptomycin

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 30 days after infusion
  A standard 3+3 trial design will be used for Welgenaleucel (UWC19) dose escalation cohorts.The dosing of Welgenaleucel (UWC19) will be divided into 5 cohorts, the subjects will receive Welgenaleucel (UWC19) once on day 14-18 after apheresis.
Dose Limiting Toxicities (DLT) | 30 days after infusion
  The 3+3 design entails that if one patient out of the first three patients has a DLT, up to three additional patients will be entered at that dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Liang Ho, MD, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan